CLINICAL TRIAL: NCT07229222
Title: Decidual-Sparing Two-Layered Simple Interrupted Myometrial Suturing With Visceral Peritoneal Closure Reduces Uterine Niche Formation After Primary Cesarean Section: A Randomized Controlled Trial
Brief Title: A Two-Layered Simple Interrupted Myometrial Suturing Reduces Uterine Niche Formation After Primary Cesarean Section
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Latif Ahmed Alnezamy, Lecturer of Obstetrics and Gynecology, Faculty of Medicine, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RC13-2-2025
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cesarean Section Complications; Scar Niche; Myometrial Remodeling; Suture Techniques
Keywords: Uterine niche; Myometrial closure; Residual myometrial thickness; Randomized controlled trial; Cesarean scar disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two-layered simple interrupted suturing of the myometrium (Active Comparator): Two-layered simple interrupted suturing of the myometrium, sparing the decidua, with closure of the visceral uterine peritoneum.
  Interventions: Procedure: Primary Cesarean Section with two-layered simple interrupted suturing of the myometrium; Diagnostic Test: Saline-infusion Sonohysterography
- Double-layered continuous suturing of the myometrium. (Active Comparator): Double-layered continuous suturing of the myometrium, sparing the decidua, with closure of the visceral uterine peritoneum.
  Interventions: Procedure: Primary Cesarean Section with double-layered continuous suturing of the myometrium; Diagnostic Test: Saline-infusion Sonohysterography

INTERVENTIONS:
Procedure: Primary Cesarean Section with two-layered simple interrupted suturing of the myometrium — All steps of cesarean section were standardized for both arms except for the type of myometrial suturing where two-layered simple interrupted suturing of the myometrium was applied.
  Arms: Two-layered simple interrupted suturing of the myometrium
Procedure: Primary Cesarean Section with double-layered continuous suturing of the myometrium — All steps of cesarean section were standardized for both arms except for the type of myometrial suturing where double-layered continuous suturing of the myometrium was applied.
  Arms: Double-layered continuous suturing of the myometrium.
Diagnostic Test: Saline-infusion Sonohysterography — At 6 months postpartum, all patients were evaluated by a single blinded sonographer experienced in niche assessment. First, transvaginal ultrasound was performed to exclude pregnancy or pelvic pathology, followed by saline-infusion sonohysterography (2D, sagittal and coronal views). A niche was defined as ≥ 2 mm myometrial indentation at the scar site. Niche depth, length, width, and residual myometrial thickness were recorded.

SUMMARY:
The purpose of the study is to determine whether two-layered simple interrupted myometrial suturing is superior to double-layered continuous suturing for the prevention of uterine niche formation after primary cesarean section.

DETAILED DESCRIPTION:
All primigravidae at or beyond 28 weeks' gestation undergoing primary cesarean section for any indication were assessed for eligibility. All participants provided written informed consent before enrolment. All patients received preoperative antibiotic prophylaxis at induction of anesthesia and postoperative prophylaxis for 24 h. A single intramuscular dose of oxytocin 10 IU was administered during the first 24 h postpartum. After confirming eligibility and obtaining consent, a trained nurse selected an envelope for each patient and revealed the allocation to the operating obstetrician. Patients were blinded to group allocation.

* Study Group: Two-layered simple interrupted suturing of the myometrium, sparing the decidua, with closure of the visceral uterine peritoneum.
* Control Group: Double-layered continuous suturing of the myometrium, sparing the decidua, with closure of the visceral uterine peritoneum.

The parietal peritoneum was left open in all cases. Hemostasis was ensured, and the number of additional hemostatic sutures was recorded. A braided polyglycolic acid 0-1 suture was used in all cases. All other steps of cesarean section were standardized.

At 6 months postpartum, all patients were evaluated by a single blinded sonographer experienced in niche assessment. First, transvaginal ultrasound was performed to exclude pregnancy or pelvic pathology, followed by saline-infusion sonohysterography (2D, sagittal and coronal views). A niche was defined as ≥ 2 mm myometrial indentation at the scar site. Niche depth, length, width, and residual myometrial thickness were recorded.

Menstrual history was obtained by an independent obstetrician/gynecologist, documenting spotting days, total bleeding days, amenorrhea, and contraceptive use.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance to participate and willingness to attend follow-up for 6 months postpartum.
* No plans for pregnancy within the follow-up period.

Exclusion Criteria:

* Known Müllerian anomalies or uterine fibroids.
* Previous uterine surgery.
* Multiple gestation.
* Chorioamnionitis, placenta previa, or placental abruption.
* Preeclampsia/eclampsia.
* Hepatic or renal dysfunction, uncontrolled diabetes, or systemic disease.
* Peripartum hemoglobin < 10 g/dL.
* Chronic corticosteroid use or smoking.
* Inability to provide consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 380 (Actual)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of uterine niche formation after primary cesarean section. | At 6 months postpartum
  Using saline-infusion sonohysterography (2D, sagittal and coronal views), a niche was defined as ≥ 2 mm myometrial indentation at the scar site.

SECONDARY OUTCOMES:
Uterine niche measurements | At 6 months postpartum
  Using saline-infusion sonohysterography (2D, sagittal and coronal views),niche depth, length, width, and residual myometrial thickness are to be recorded.
Total operative time. | Intraoperative
  The operation room nurse recorded the time lapse between the skin incision and the end of skin suturing.
The correlation between niche width and menstrual cycle abnormalities. | At 6 months postpartum
  For participants diagnosed with uterine niche, menstrual history was obtained by an independent obstetrician/gynecologist, documenting spotting days, total bleeding days, amenorrhea, and contraceptive use.
The association between active labour at the time of cesarean and niche formation. | Cervical dilatation was evaluated immediately preoperative, while the association was evaluated at 6 months postpartum
  Active labour in primigravida was identified when the cervical dilatation is equal to or more than 3 cm.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED ALNEZAMY, MD, Principal Investigator — Lecturer of Obstetrics and Gynecology, Faculty of Medicine, Benha University
Locations (1):
- Benha Univesity Hospital, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jordans IPM, de Leeuw RA, Stegwee SI, Amso NN, Barri-Soldevila PN, van den Bosch T, Bourne T, Brolmann HAM, Donnez O, Dueholm M, Hehenkamp WJK, Jastrow N, Jurkovic D, Mashiach R, Naji O, Streuli I, Timmerman D, van der Voet LF, Huirne JAF. Sonographic examination of uterine niche in non-pregnant women: a modified Delphi procedure. Ultrasound Obstet Gynecol. 2019 Jan;53(1):107-115. doi: 10.1002/uog.19049. PMID 29536581
- [Background] Monteagudo A, Carreno C, Timor-Tritsch IE. Saline infusion sonohysterography in nonpregnant women with previous cesarean delivery: the "niche" in the scar. J Ultrasound Med. 2001 Oct;20(10):1105-15. doi: 10.7863/jum.2001.20.10.1105. PMID 11587017
- [Background] Klein Meuleman SJM, Min N, Hehenkamp WJK, Post Uiterweer ED, Huirne JAF, de Leeuw RA. The definition, diagnosis, and symptoms of the uterine niche - A systematic review. Best Pract Res Clin Obstet Gynaecol. 2023 Aug;90:102390. doi: 10.1016/j.bpobgyn.2023.102390. Epub 2023 Jul 15. PMID 37506497
- [Background] Vervoort A, Vissers J, Hehenkamp W, Brolmann H, Huirne J. The effect of laparoscopic resection of large niches in the uterine caesarean scar on symptoms, ultrasound findings and quality of life: a prospective cohort study. BJOG. 2018 Feb;125(3):317-325. doi: 10.1111/1471-0528.14822. Epub 2017 Aug 28. PMID 28703935
- [Background] Vikhareva Osser O, Valentin L. Clinical importance of appearance of cesarean hysterotomy scar at transvaginal ultrasonography in nonpregnant women. Obstet Gynecol. 2011 Mar;117(3):525-532. doi: 10.1097/AOG.0b013e318209abf0. PMID 21343754
- [Background] Baranov A, Gunnarsson G, Salvesen KA, Isberg PE, Vikhareva O. Assessment of Cesarean hysterotomy scar in non-pregnant women: reliability of transvaginal sonography with and without contrast enhancement. Ultrasound Obstet Gynecol. 2016 Apr;47(4):499-505. doi: 10.1002/uog.14833. Epub 2016 Feb 29. PMID 25720922
- [Result] Osser OV, Jokubkiene L, Valentin L. Cesarean section scar defects: agreement between transvaginal sonographic findings with and without saline contrast enhancement. Ultrasound Obstet Gynecol. 2010 Jan;35(1):75-83. doi: 10.1002/uog.7496. PMID 20034000
- [Result] Antoine C, Meyer JA, Silverstein JS, Alexander J, Oh C, Timor-Tritsch IE. The Impact of Uterine Incision Closure Techniques on Post-cesarean Delivery Niche Formation and Size: Sonohysterographic Examination of Nonpregnant Women. J Ultrasound Med. 2022 Jul;41(7):1763-1771. doi: 10.1002/jum.15859. Epub 2021 Nov 2. PMID 34726789
- [Result] Tsuji S, Katsura D, Tokoro S, Inatomi A, Nobuta Y, Yoneoka Y, Amano T, Murakami T. Two-layer interrupted versus two-layer continuous sutures for preventing cesarean scar defect: a randomized controlled trial. BMC Pregnancy Childbirth. 2025 Mar 7;25(1):248. doi: 10.1186/s12884-025-07353-1. PMID 40055610